CLINICAL TRIAL: NCT04688216
Title: Developing the Best Risk Assessment System of Multidrug-resistant Organisms Infection in Critically Ill Patients Based on Big Data Analysis Technology
Brief Title: Developing a Risk Assessment System of Multidrug-resistant Organisms Infection
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-408
Record Dates: First submitted 2020-12-06; First posted 2020-12-29 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2022-12

CONDITIONS: Bacterial Infections
Keywords: risk assessment system; multidrug-resistant organisms; ICU
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MDRO
  Interventions: Other: risk factors of infection with multidrug-resistant organisms
- Non-MDRO
  Interventions: Other: risk factors of infection with multidrug-resistant organisms

INTERVENTIONS:
Other: risk factors of infection with multidrug-resistant organisms — 1. General information: age, gender, length of stay in ICU, method of admission, tubes taken at the time of admission, APACHEⅡ score, surgery, laboratory tests (PCT, CRP, WBC), pressure sores, etc.
  2. Iatrogenic factors: days of using ventilator, days of using antibacterial drugs, types of antibacterial drugs, use of glucocorticoids, use of immunosuppressants, days of central venous intubation, days of indwelling catheters, days of arterial catheterization, and other indwelling catheters.
  3. The patient's own related factors: diagnosis, whether complicated with hypertension or diabetes; whether exist malignant tumor, primary lung infection, hypoproteinemia; whether antibiotic treatment before admission; fever and fever days, whether diarrhea occurs

SUMMARY:
1. A retrospective analysis was performed to determine the prevalence of multidrug- resistant organisms infection in ICU from October 2017 to October 2019.
2. Non-MDRO patients were selected by random sampling in a ratio of 1:1 to the final MDRO group during the same period , and select the risk factors of infection with multi-drug resistant bacteria by comparing the two groups.
3. Randomly select 30% of the sample size as the validation set, and the remaining 70% for the training set to establish a model. Using multi-factor Logistic regression, decision tree classification, artificial neural network, support vector machine, Bayesian network Method to establish risk assessment system for multidrug-resistant organisms infection respectively.Using validation set data to calculate the area under the ROC curve (AUC) and sensitivity, specificity of models and comparing the prediction accuracy of several models. Finally, choose a more suitable risk assessment system for multidrug-resistant organisms infection.
4. Predict the patient's infection risk level according to the best risk assessment system and develop a low-to-high intervention plan.

ELIGIBILITY:
Inclusion Criteria：

* Duration of ICU admission ≥ 48h
* no less than 18 years old

Exclusion Criteria:

* Patients with MDRO infection at the time of admission
* Lack of case data
* MDRO colonized patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ①Length of stay in ICU is more than 48h; ② no less than 18 years old.
Sampling Method: Probability Sample
Enrollment: 917 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
multidrug-resistant organisms infection | From date of ICU admissions until the date of ICU discharge or date of diagnosis of multidrug-resistant organisms infection , whichever came first, assessed up to 24 months
  Ratio of the number of multi-drug resistant bacterial infections to the total number of patients

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided